CLINICAL TRIAL: NCT04842305
Title: Induction of SARS-CoV-2 Spike Glycoprotein Antibodies in Saliva and Plasma in Response to a COVID-19 Infection, Systemic COVID-19 Vaccination, and the Combination of COVID-19 and Vaccination
Brief Title: Mucosal Immunity in Terms of SARS-CoV-2 Antibodies in Saliva After COVID-19 Infection and Vaccination
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lenanrt Friis-Hansen (Other)
Responsible Party: Sponsor-Investigator, Lenanrt Friis-Hansen, Department of Clinical Biochemistry MD, DMSc, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Other Study IDs: P-2021-224
Record Dates: First submitted 2021-04-05; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: sars-cov-2 antibodies; saliva; mucosal immunity; vaccination; covid19; spike glycoprotein
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- G1: Control group: SARS-CoV-2 naïve persons who have neither been vaccinated nor have had COVID-19 (controls)
  Interventions: Diagnostic Test: Blood- and saliva tests
- G2: COVID-19 infected: Persons who have had COVID-19
  Interventions: Diagnostic Test: Blood- and saliva tests
- G3: COVID-19 vaccinated: Persons who have been vaccinated with Pfizer-BioNTech BNT162b2, Moderna mRNA-1273 or AstraZeneca ChAdOx1-S
  Interventions: Diagnostic Test: Blood- and saliva tests
- G4: COVID-19 infected and vaccinated: Individuals who have been infected with COVID-19 and subsequently been vaccinated
  Interventions: Diagnostic Test: Blood- and saliva tests

INTERVENTIONS:
Diagnostic Test: Blood- and saliva tests — Measurement of SARS-CoV-2 spike glycoprotein RBD antibodies in plasma and saliva

SUMMARY:
The Primary Objective of This Single-center Study is to Investigate the SARS-CoV-2 Spike Glycoprotein RBD Antibody Concentration in Saliva and Serum in Healthy Non Vaccinated and Non-SARS-CoV-2 Infected, COVID-19 Convalescents, Persons Vaccinated With Pfizer-BioNTech BNT162b2, Moderna mRNA-1273 or AstraZeneca ChAdOx1 nCov-19 AZD1222 Vaccines, and Convalescent COVID-19 Patients That Have Subsequently Been Vaccinated. A Potential Difference in the Immunoglobulin Concentrations of the Pfizer-BioNTech BNT162b2 Vaccine, Moderna mRNA-1273 vaccine and the AstraZeneca ChAdOx1-S Vaccine Will be Uncovered. This Knowledge About the Mucosal Immunity Will be Important for Further Designing of Vaccine Strategies.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Both Hospital staff as well as non-health care workers will be invited to participate

Exclusion Criteria:

* Individuals not fulfilling the inclusion criteria or declining blood or saliva collection.
* Exclusion criteria are neck breathers (tracheostomy/laryngectomy patients) or other nasopharyngeal or oropharyngeal anomalies that do not allow for sampling using Salivette.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who belong to one of the following four groups will be included G1=SARS-COV-2 Naïve (=Not SARS-CoV-2 vaccinated and COVID-19 negative), G2=COVID-19 convalescents, G3=Vaccinated with Pfizer-BioNTech BNT162b2, Moderna mRNA-1273 or AstraZeneca ChAdOx1-S vaccine, G4=COVID-19 positive and vaccinated with Pfizer-BioNTech BNT162b2, Moderna mRNA-1273 or AstraZeneca ChAdOx1-S vaccine
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Titer of SARS-CoV-2 spike glycoprotein RBD antibodies in saliva and plasma | Between 21 and 200 days after infection/vaccination
  Detection of SARS-CoV-2 spike glycoprotein RBD antibodies in saliva and plasma in participants who have been infected with COVID-19, vaccinated with Pfizer-BioNTech/Moderna mRNA-1273/AstraZeneca or infected and vaccinated

SECONDARY OUTCOMES:
Titer of SARS-CoV-2 spike glycoprotein RBD antibodies in saliva and plasma | Between 21 and 200 days after vaccination
  Comparison of SARS-CoV-2 spike glycoprotein RBD antibodies (in saliva and plasma) between participants vaccinated with Pfizer-BioNTech, Moderna mRNA-1273 and AstraZeneca

IPD SHARING:
Plan to Share IPD: Undecided